CLINICAL TRIAL: NCT05367258
Title: Umbilical Endometriosis: a Comparison of Medical and Surgical Therapy and Pathogenetic Considerations
Acronym: UMBEND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Direzione Ginecologia, Professor Nicola Berlanda, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 2283
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis of Umbilicus; Endometriosis in Scar of Skin; Endometriosis-related Pain; Endometriosis
Keywords: Surgical treatment; Medical therapy; Satisfaction
MeSH Terms: conditions — Endometriosis; Personal Satisfaction | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients satisfaction after medical and surgical treatment for umbilical endometriosis — It is a retrospectively evaluation of cases of umbilical endometriosis in our clinic over the last 30 years, based on the review of medical records and on outpatient follow-up visits. The questionnaire are filled in routinely by patients attending the endometriosis center of this institute every 6 months. We will collect data relating to these questionnaires referring prospectively to the study period. If the questionnaires have not already been filled in by the patient, she will be contacted to fill them in, after signing the informed consent of the study.

SUMMARY:
Endometriosis is the presence of endometrial glands and stroma outside the uterine cavity. About 5% of women of reproductive age suffer from the disease.

The pelvis is the most frequent site of endometriotic lesion and the most common pelvic localisations are peritoneal, ovarian, and deep infiltrating endometriosis. However, endometriosis can also localize outside the pelvis, for example involving the umbilicus, omentum, appendix, liver, diaphragm, pleura and lungs, vulva, and surgical scars.

The majority of extrapelvic endometriosis implants are located in the skin, and most of them are of iatrogenic origin, following laparotomy, laparoscopic procedures, and episiotomies; only a minority of cases are of primary origin.

Umbilical endometriosis is a very rare presentation of endometriosis (0.5-1% of cases of extrapelvic endometriosis).

Pathogenetic hypotheses of primary umbilical endometriosis include: hematic or lymphatic dissemination of endometrial cells from the peritoneum to the umbilicus through obliterated umbilical arteries; migration of endometrial cells through the venous or lymphatic circulation; metaplasia of urachus remnant or release of endometrial cells that during labor and delivery may contaminate the umbilical cord emergence. Secondary umbilical endometriosis is probably due to the proliferation and subsequent dissemination of iatrogenically implanted endometrial cells in laparotomy or laparoscopic scars. In 20% of cases, umbilical endometriosis is associated with pelvic endometriosis. In these patients, it is probable that endometriotic cells may migrate from the endometriotic implants to the umbilical site.

This migration process could be favored by fascia defects at the umbilical level. In fact, reports in the literature describe cases of umbilical endometriosis coexisting with umbilical hernia.

The clinical presentation consists of an umbilical nodule of variable color (red, blue, black, flesh-colored), ranging in size from 0.5 to 3 cm.

Pathognomonic symptoms are: bleeding and/or pain in the umbilical site of catamenial type, cutaneous hyperesthesia. Catamenial symptomatology associated with the nodule, which makes the diagnosis easier, is present in only 75% of cases.

In asymptomatic cases the differential diagnosis of the nodule of umbilical endometriosis is more difficult (hernia, hematoma, cyst, dermatological disorders, tumor metastasis).

Instrumental examinations useful for differential diagnosis and definition of nodule size include soft tissue ultrasound, CT scan and MRI.

Definitive diagnosis is only by histologic examination of the tissue. Exploratory laparoscopy is not indicated unless concomitant pelvic endometriosis is suspected.

The recommended treatment of umbilical endometriosis is surgical, consisting of complete removal of the endometriosis nodule, omphalectomy, and subsequent reconstruction of the umbilicus.

Recurrence rates after surgery are around 6% at 12 months in a large Japanese court, with no difference between taking and not taking postoperative hormonal therapy, while they are reduced to almost 0% in case of resection including a large portion of peritoneum.

Medical therapy, on the other hand, alleviates the associated algic symptoms by reducing the size of the nodule.

There are very few data on the efficacy of medical therapy; in a study with a very small number of cases an efficacy of 91.7% with dienogest and 51.1% with estroprogestinic pill is reported. There are no studies comparing medical and surgical therapy for the treatment of umbilical endometriosis.

Radical excision is recommended to avoid local recurrences and to avoid the risk of malignant transformation, although it is extremely rare (only 2 cases reported).

In literature, spontaneous resolution has been described in only one pregnant woman.

To date, few studies have evaluated umbilical endometriosis. Moreover, no study has ever formally compared the long-term efficacy of surgical or medical therapy for umbilical endometriosis.

This is a observational, retrospective/prospective and monocentric study; it is based on the review of medical records and on outpatient follow-up visits of patients in our clinic with umbilical endometriosis from 1990.

The principal aim of the study is to evaluate the effectiveness of medical and surgical treatments in terms of satisfaction, psychological state, health-related quality of life of patients suffering from this clinical condition. Moreover, global patient's condition and severity of the patient's symptoms are evaluated The secondary aim is to investigate the pathogenetic aspects of this clinical condition.

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometrial glands and stroma outside the uterine cavity. About 5% of women of reproductive age suffer from the disease.

The pelvis is the most frequent site of endometriotic lesion and three types of pelvic endometriosis can be clinically distinguished: peritoneal, ovarian, and deep infiltrating endometriosis.

However, endometriosis can also localize outside the pelvis: extra-pelvic foci may be found involving the umbilicus, omentum, appendix, liver, diaphragm, pleura and lungs, vulva, and surgical scars.

The majority of extrapelvic endometriosis implants are located in the skin, and most of them are of iatrogenic origin, following laparotomy, laparoscopic procedures, and episiotomies; only a minority of cases are of primary origin.

Umbilical endometriosis - first described by Villar in 1886 - is a very rare presentation of endometriosis, with a prevalence ranging from 0.5-1% of cases of extrapelvic endometriosis The proliferation and subsequent dissemination of iatrogenically implanted endometrial cells in laparotomy or laparoscopic scars would seem to be the cause of the occurrence of secondary umbilical endometriosis. Obviously this is not true in cases of primary umbilical endometriosis, in which case the pathogenic hypotheses include: hematic or lymphatic dissemination of endometrial cells from the peritoneum to the umbilicus through obliterated umbilical arteries; migration of endometrial cells through the venous or lymphatic circulation; metaplasia of urachus remnant or release of endometrial cells that during labor and delivery may contaminate the umbilical cord emergence. In 20% of cases, umbilical endometriosis is associated with pelvic endometriosis. In these patients, it is possible to speculate that endometriotic cells may migrate from the endometriotic implants to the umbilical site.

This migration process could be favored by fascia defects at the umbilical level. In fact, cases of umbilical endometriosis coexisting with umbilical hernia are described in the literature.

The clinical presentation consists of an umbilical nodule of variable color (red, blue, black, flesh-colored), ranging in size from 0.5 to 3 cm.

Pathognomonic symptoms are: bleeding and/or pain in the umbilical site of catamenial type, cutaneous hyperesthesia. Catamenial symptomatology associated with the nodule, which makes the diagnosis easier, is present in only 75% of cases.

In asymptomatic cases the nodule of umbilical endometriosis should be differentially diagnosed with hernia, hematoma or cyst and with some dermatological disorders such as pyogenic granuloma, umbilical polyp, melanocytic nevus, seborrheic keratosis, epithelial inclusion cysts, desmoid tumor, hemangioma and granular cell tumor. Furthermore, it should be ruled out that it is not a Sister Joseph's nodule, a sentinel of tumor metastasis, whose clinical symptomatology is similar to umbilical endometriosis, although the nodule tends to be more irregular and the symptoms non-cyclic. A case of umbilical metastasis from endometrial carcinoma, synchronous with umbilical endometriosis, is reported.

Instrumental examinations useful for differential diagnosis and definition of nodule size include soft tissue ultrasound, CT scan, and MRI.

Definitive diagnosis is provided only by histologic examination of the tissue. Exploratory laparoscopy is not indicated unless concomitant pelvic endometriosis is suspected.

The recommended treatment of umbilical endometriosis is surgical, consisting of complete removal of the endometriosis nodule, omphalectomy, and subsequent reconstruction of the umbilicus.

Recurrence rates after surgery are around 6% at 12 months in a large Japanese court, with no difference between taking and not taking postoperative hormonal therapy, while they are reduced to almost 0% in case of resection including a large portion of peritoneum.

Medical therapy, on the other hand, alleviates the associated algic symptoms by reducing the size of the nodule.

In the literature there are very few data on the efficacy of medical therapy; in a study with a very small number of cases an efficacy of 91.7% with dienogest and 51.1% with estroprogestinic pill is reported. There are no studies comparing medical and surgical therapy for the treatment of umbilical endometriosis.

Radical excision is recommended to avoid local recurrences and to avoid the risk of malignant transformation, although it is extremely rare (only 2 cases reported in the literature).

In literature, spontaneous resolution has been described in only one pregnant woman.

To date, there are few studies in the literature that have evaluated umbilical endometriosis.

Moreover, no study has ever formally compared the long-term efficacy of surgical or medical therapy for umbilical endometriosis.

This is an observational, retrospective/prospective and monocentric study; it is based on the review of medical records and on outpatient follow-up visits of patients in our clinic with umbilical endometriosis. This is a study design that it is best suited to a low prevalence of disease.

The principal aim of the study is the assessment of umbilical endometriosis cases in our clinic over the last 30 years in order to evaluate the effectiveness of medical and surgical treatments in terms of satisfaction, psychological state, health-related quality of life of patients suffering from this clinical condition. Moreover, global patient's condition and severity of the patient's symptoms are evaluated.

The secondary aim is to investigate the pathogenetic aspects of this clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-50 years with a diagnosis of umbilical endometriosis, in the presence or absence of other endometriotic localizations, referred to our tertiary-care endometriosis center " Fondazione IRCCS Ospedale Maggiore Policlinico", Milan, from 1 January 1990 to 01 March 2022.

Exclusion Criteria:

* Exclusion criteria are the presence of concomitant psychiatric disease, chronic intestinal disease (Chron's disease or ulcerative rectocolitis), or disease that may cause pelvic pain (e.g., pelvic venous varices and salpingitis outcomes).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the patients referred to our endometriosis clinic and/or underwent surgery from 1 January 1990 to 01 March 2022 with a diagnosis of umbilical endometriosis were selected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Degree of patient satisfaction | 30 years
  a five-level Likert scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied and very dissatisfied) to evaluate the effectiveness of medical and surgical treatments for umbilical endometriosis.
The patient's global condition | 30 years
  Patients' Global Impression of Change (PGIC) scale, a composed of seven levels (greatly improved, much improved, minimally improved, unchanged, minimally worsened, very worsened, greatly worsened) to evaluate the effectiveness of medical and surgical treatments for umbilical endometriosis.
Severity of symptoms | 30 years
  Patients' Global Impression of Severity (PGIS) scale, a scale consisting of five levels (none, mild, moderate, severe, very severe)
HADS- Hospital Anxiety and Depression Scale | 30 years
  The HADS questionnaire is a self-assessment mood scale specifically designed for use in non-psychiatric hospital outpatients to determine states of anxiety and depression. It comprises 14 questions, 7 for the anxiety subscale and 7 for the depression subscale.
The Short Form Survey, SF-12 | 30 years
  The SF-12 health survey, developed from the original SF-36 questionnaire, is a well-known, validated, selfadministered 12-item instrument. It measures health dimensions covering functional status, well-being, and overall health. Information from the 12 items is used to construct Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) measures, with higher scores indicating better health perception.

SECONDARY OUTCOMES:
Pathogenetic aspects | 30 years
  Study of the pathogenesis on a case-by-case basis depending on the patient's previous physiological and pathological medical history.
Comparison between medical and surgical therapy | 30 years
  Comparison through the degree of patient satisfaction, evaluated with Likert scale (used for 1st primary outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy